CLINICAL TRIAL: NCT07178808
Title: PHASE II EVALUATION OF CYTOREDUCTION SURGERY AND HYPERTHERMIC INTRAPERITONEAL CHEMOTHERAPY (CRS/HIPEC) IN GASTRIC CANCER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Banner Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1480-262
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (Experimental): Patients will undergo cytoreduction & hyperthermic intraperitoneal chemotherapy
  Interventions: Procedure: Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy

INTERVENTIONS:
Procedure: Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy — CRS/HIPEC involves aggressive surgical cytoreduction of all visible and palpable tumors, followed by the synergistic use of heated and high dose chemotherapy to address microscopic residual disease.

SUMMARY:
This is a Phase II treatment study analyzing the role of preoperative chemotherapy, preoperative laparoscopic HIPEC, and gastrectomy with CRS/HIPEC in gastric adenocarcinoma patients with cytology-positive only carcinomatosis, radiologically-occult carcinomatosis, or radiology apparent peritoneal-surface only metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18 years and above. There will be no upper age restriction. 2)ECOG performance status ≤ 2. (See Appendix A -ECOG Performance Status Scale). 3)Cytologic or histologic proof of adenocarcinoma of the stomach or gastroesophageal junction.

  4)Adequate renal, and bone marrow function:
  1. Leukocytes >= 3,000/uL
  2. Absolute neutrophil count >= 1,500/uL
  3. Platelets >= 60,000/Ul
  4. Serum creatinine <= 1.5 mg/dL 5)Distant metastatic disease of peritoneum may be visualized on imaging:

  <!-- -->

  1. Positive peritoneal cytology only
  2. Carcinomatosis on diagnostic laparoscopy or laparotomy.

     Exclusion Criteria:
* 1)Distant metastatic disease not limited to peritoneum:

  1. Solid organ metastases (liver, central nervous system, lung). 2) Infections such as pneumonia or wound infections that would preclude protocol therapy.

     3) Women with a positive urine or serum pregnancy test are excluded from this study; women ofchildbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to refrain from breast feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence.

     4)Participants with unstable angina or New York Heart Association Grade II or greater congestive heart failure.

     5) Participants deemed unable to comply with study and/or follow-up procedures. 6)Participants with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2031-02-22 (Estimated)

PRIMARY OUTCOMES:
To assess improvements in survival in gastric adenocarcinoma patients with occult or apparent carcinomatosis after cytoreductive surgery and hyperthermic intraperitoneal chemotherapy | From enrollment up to 60 months
  To determine if preoperative laparoscopic HIPEC and chemotherapy followed by cytoreductive surgery (CRS), gastrectomy and HIPEC in patients with peritoneal surface-only metastasis will improve PFS and/or OS from date of diagnosis of metastatic gastric adenocarcinoma

SECONDARY OUTCOMES:
To study recurrence pattern in patients with recurrence during the study period | From enrollment up to 60 months
  Patterns of tumor recurrence and survival will be assessed by reviewing routine surveillance imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Banner MD Anderson Cancer Center, Gilbert, Arizona, United States

IPD SHARING:
Plan to Share IPD: No